CLINICAL TRIAL: NCT01770262
Title: Development of Non-invasive Method for Quantifying Vitamin D Levels in the Body Using Spectroscopy
Status: Withdrawn | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Ruppin Acdemic Center (Other)
Responsible Party: Sponsor
Other Study IDs: DVitamin-HMO-CTIL
Record Dates: First submitted 2013-01-13; First posted 2013-01-17 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2012-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples for quantification of vitamin D levels

GROUPS / COHORTS (2):
- Osteoporosis: Hospitalized subjects diagnosed with osteoporosis
- Healthy

SUMMARY:
Lack in vitamin D reduces the absorption of calcium in the body, accelerates bone loss and may increase the risk of fractures due to osteoporosis. An algorithm that will allow immediate and non-invasive quantification of vitamin D levels will shorten the time of diagnosis, reduce lab costs and prevent hazards or discomfort to the patient associated with a blood test.

The goal of the study is therefore to develop a non-invasive method for quantifying vitamin D levels in the body using spectroscopy.

40 subjects will be recruited: 20 hospitalized patients in the rehabilitation department, diagnosed with osteoporosis and 20 healthy subjects. Spectroscopy will be used with visible light on the subject's skin and middle infrared (MIR) on the blood sample to find correlation with the chemical lab test results.

DETAILED DESCRIPTION:
Lack in vitamin D reduces the absorption of calcium in the body, accelerates bone loss and may increase the risk of fractures due to osteoporosis. Vitamin D can be ingested by foods and specific supplements, but the main source for the vitamin is its synthesis in the skin by using sun radiation. Today, quantification of vitamin D levels is performed using a blood test. Mostly, the physician will send the patient to check the levels and vitamin D if he suffers from osteoporosis, hypertension, renal impairment, suspected for activity of the thyroid gland, tuberculosis or sarcoidosis.

Studies have shown that it is possible to quantify the different elements in the contents of the blood, such as melanin and hemoglobin, using spectroscopy of the skin (Zonios et al, 2001; Tseng et al, 2009), but to the investigators' knowledge, the identification of levels and vitamin D in similar means has not been reported in professional literature.

The rationale for this research: an algorithm that will allow immediate and non-invasive quantification of vitamin D levels will shorten the time of diagnosis, reduce lab costs and prevent hazards or discomfort to the patient associated with a blood test.

The goal of this study is therefore to develop a non-invasive method for quantifying vitamin D levels in the body using spectroscopy.

Methods:

40 subjects aged 18-65 will be recruited for this research: 20 patients be recruited from the population of patients in the rehabilitation department who were diagnosed with osteoporosis. Also, 20 healthy subjects will be recruited.

All participants will be able to understand the study protocol and sign a consent form independently.

In this study, the investigators will look for a correlation between the results of conventional blood test for detection of vitamin D levels in the blood and the results of measurements of spectral examinations that will be performed on various locations on the upper body of the subject. These measurements will take place in Hillel Yaffe Medical Center as the subject arrives to the chemistry lab for the blood test. Visible light spectrometer (manufactured by Ocean Optics, USB 2000 model), connected to an optical fiber (manufactured by Ocean Optics, diameter 1mm) will be used. The measurement will use a light source (Fiberoptics Technology Inc. company., Model SOL-R 150) connected also to an optical fiber. Both ends of the fiber will be positioned on the upper body of the patient one of two configurations: for areas with greater thickness, e.g. the forearm, the fibers would be placed next to each other on the same side of the limb to measure the return of the light, and in areas with smaller tissue thickness, e.g. finger tip, the fibers will be placed to both sides of an organ and record light transmission through the target.

First, the investigators will attempt to find correlation between the spectral analysis results of the visible wavelengths and the blood test. Then the investigators will further compare the subjects' blood samples using FTIR spectrometer in the mid infrared (device manufactured by Oriel, Model MIR8025). The device is equipped with plug-ATR (Attenuated Total Reflectance) and allows testing of a small sample of fluids. Vials of samples delivered to Rupin on foil-wrapped test using a cooler with ice will be tested in Ruppin on the day of extraction. The samples will be disposed of as biological waste.

Trial protocol:

Each subject will arrive at the lab at Hillel Yaffe Medical Center. the subject will read and sign an informed consent form for participation in the study. The subject will fill out a short questionnaire reporting on the nature of sun exposure, dietary habits and chronic medications.

Then two tests will be performed:

1. Blood test for vitamin D levels.
2. Test using the spectrometer: two fiber optic guided by the researchers on different places on the torso of the patient, when one side of the fiber optic is connected to a light source and the anther optical fiber end is connected to the spectrometer.

There is no expected risk or discomfort to the subject beyond the risk associated with regular blood tests.

Spectral test to be held Ruppin on the patient's blood samples, as described in the methods, and will not require the presence of the patient.

Data analysis:

Several algorithms will be developed to be used on the spectral database, in order to identify individuals suffering from vitamin D deficiency.

The data processing will be as follows:

1. Statistical analyzes will be carried out using regression methods to find correlation between the level of vitamin D quantified with laboratory chemical test of the blood and spectral measurements in the visible light as performed at the hospital in different areas of the body.
2. Statistical analyzes will be carried out using regression methods to find correlation between the level of vitamin D quantified with laboratory chemical test of the blood and spectral measurements in middle infrared (MIR), as performed on blood samples taken from subjects.
3. The tested population will be divided into two groups according to the blood test results: subjects defined as having vitamin D deficiency and subjects classified as having normal vitamin D levels. Clustering methods of analysis will be carried out, such as PCA and LDA, to find distinguishing characteristic between the two populations.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Pregnant
* Cannot understand or sign a consent form independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 subjects aged 18 years and above will be recruited for this research: 20 patients be recruited from the population of patients in the rehabilitation department who were diagnosed with osteoporosis. Also, we will recruit 20 healthy subjects.
  All participants will be able to understand the study protocol and sign a consent form independently.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Vitamin D levels | At baseline
  No followup will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Mordechi Hallak, MD, MPA, Principal Investigator — Hillel Yaffe Medical Center; Sigal Portnoy, PhD, Study Director — Hadassah Medical Organization; ben zion Dekel, PhD, Study Director — Rupin academic center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel